CLINICAL TRIAL: NCT00005717
Title: Medication Adherence in COPD--A Self-Regulation Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4926; R01HL042489 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-06

CONDITIONS: Lung Diseases, Obstructive; Bronchitis; Emphysema; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive; Bronchitis; Emphysema; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To test the effectiveness of a self-management program for chronic obstructive disease (COPD) patients. The program to improve adherence could be conducted by nurses or other clinic staff in settings where comprehensive rehabilitation services were not available.

DETAILED DESCRIPTION:
BACKGROUND:

In 1990, the available data on medication adherence among chronic obstructive pulmonary disease (COPD) patients consistently indicated that adherence was a significant problem. This was a particularly distressing finding, considering that pharmacological therapy was considered the backbone of COPD management in settings where comprehensive rehabilitation services were limited. Despite the importance of this issue and a large data base on how to enhance medication adherence among medical populations, there had been no empirical investigations evaluating the implementation of these strategies with COPD patients.

DESIGN NARRATIVE:

The prospective, controlled study randomized 230 emphysema and chronic bronchitis patients from an urban university medical center into either a "usual care", control group or into a self-management skills training program for improving adherence. The training program was based on self-management procedures for enhancing adherence which had proven efficacious with diverse populations.

Self-reported and objective measures of adherence were examined during the two month baseline period and the one year follow-up in the controlled study. A range of possible covariates including demographics, patient characteristics, treatment, and therapeutic outcome variables were also collected during the baseline phase and at the 6-month and 12-month follow-up visits in the controlled study to evaluate their relationship to the observed adherence levels.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-08; Study Completion 1995-07 (Actual)